CLINICAL TRIAL: NCT05710874
Title: A Prospective, Randomized, Clinical Study on the Effects of Casein Phosphopeptide Amorphous Calcium Phosphate Paste, Fluoride and a Combination on the Evolution of White Spot Lesions in Orthodontic Patients After Debonding.
Brief Title: A Prospective, Randomized, Clinical Study on the Effects of CPP-ACP-paste, Fluoride and a Combination on the Evolution of White Spot Lesions in Orthodontic Patients After Debonding.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BC-01938
Record Dates: First submitted 2023-01-11; First posted 2023-02-02 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: White Spot Lesion; Orthodontic Appliance Complication
Keywords: orthodontics; orthodontic brackets; dental caries; decalcification; caseins; fluorides
MeSH Terms: conditions — Dental Caries | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CPP-ACP paste (Experimental): Daily application of CPP-ACP (Casein phosphopeptide amorphous calcium phosphate) paste (Tooth Mousse®) in addition to twice daily use of conventional toothpaste.
  Interventions: Other: CPP-ACP paste
- CPP-ACPF paste (Experimental): Daily application of CPP-ACPF (Casein phosphopeptide amorphous calcium phosphate in combination with fluoride) paste (MI Paste Plus®) in addition to twice daily use of conventional toothpaste..
  Interventions: Other: CPP-ACPF paste
- 1.25% fluoride gel (Experimental): Weekly application of 1.25% fluoride gel (Elmex Medical Gel®) in addition to twice daily use of conventional toothpaste.
  Interventions: Other: 1.25% fluoride gel
- Conventional (Placebo Comparator): Twice daily use of conventional toothpaste.
  Interventions: Other: Conventional

INTERVENTIONS:
Other: CPP-ACP paste — Daily application of CPP-ACP (Casein phosphopeptide amorphous calcium phosphate) paste (Tooth Mousse®) in addition to twice daily use of conventional toothpaste.
  Arms: CPP-ACP paste
Other: CPP-ACPF paste — Daily application of CPP-ACPF (Casein phosphopeptide amorphous calcium phosphate in combination with fluoridepaste) (MI Paste Plus®) in addition to twice daily use of conventional toothpaste.
  Arms: CPP-ACPF paste
Other: 1.25% fluoride gel — Weekly application of 1.25% fluoride gel (Elmex Medical Gel®) in addition to twice daily use of conventional toothpaste.
  Arms: 1.25% fluoride gel
Other: Conventional — Twice daily use of conventional toothpaste.
  Arms: Conventional

SUMMARY:
The goal of this randomized clinical trial is to compare the influence of casein phosphopeptide amorphous calcium phosphate (CPP-ACP), CPP-ACP in combination with fluoride (CPP-ACPF), high fluoride concentration, and conventional fluoride toothpaste on the color and size of white spot lesions (WSLs) in orthodontic patients following bracket removal.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with fixed orthodontic appliances at the Ghent University Hospital who developed at least three WSLs at debonding were included. Informed consent had to be obtained from the patient, both verbally and written.

Exclusion Criteria:

* Patients were excluded from the study if enamel demineralization was already present before orthodontic treatment.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 107 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Evolution of the relative area of the white spot lesions | The change in relative area between the end of orthodontic treatment (T0) and 2 months after the end of orthodontic treatment (T1) is measured.
  ImageJ® (National Institutes of Health, Bethesda, MD, USA) was used to measure the relative area. In order to measure the relative area of the white spot lesions, the affected tooth was trimmed out of the original photo and the entire buccal surface was measured in absolute pixels. After this, the white spot lesion was outlined and measured in pixels.
Evolution of the relative area of the white spot lesions | The change in relative area between the end of orthodontic treatment (T0) and 4 months after the end of orthodontic treatment (T2) is measured. Patients participate in the study for 4 months.
  ImageJ® (National Institutes of Health, Bethesda, MD, USA) was used to measure the relative area. In order to measure the relative area of the white spot lesions, the affected tooth was trimmed out of the original photo and the entire buccal surface was measured in absolute pixels. After this, the white spot lesion was outlined and measured in pixels.
Evolution of the Andersson Index of the white spot lesions | The change in Andersson Index between the end of orthodontic treatment (T0) and 2 months after the end of orthodontic treatment (T1) is measured.
  The Andersson Index (AI) was determined on the basis of the clinical pictures.
Evolution of the Andersson Index of the white spot lesions | The change in Andersson Index between the end of orthodontic treatment (T0) and 4 months after the end of orthodontic treatment (T2) is measured. Patients participate in the study for 4 months.
  The Andersson Index (AI) was determined on the basis of the clinical pictures.

SECONDARY OUTCOMES:
Gingival Index | The Gingival Indexis measured at the end of orthodontic treatment (T0), at 2 months after the end of orthodontic treatment (T1) and at 4 months after the end of orthodontic treatment (T2). Patients participate in the study for 4 months.
  The Gingival Index is determined by the maximum score measured on the included teeth. Score 0 means no gingival inflammation and score 1 means gingival inflammation.
Plaque Index | The Plaque Index is measured at the end of orthodontic treatment (T0), at 2 months after the end of orthodontic treatment (T1) and at 4 months after the end of orthodontic treatment (T2). Patients participate in the study for 4 months.
  The Gingival Index is determined by the maximum score measured on the included teeth. Score 0 means no plaque and score 1 means plaque.
Patient's use of the tooth paste | The patient's use of the tooth paste is determined at 2 months after the end of orthodontic treatment (T1) and at 4 months after the end of orthodontic treatment (T2). Patients participate in the study for 4 months.
  According to the patient's use of toothpaste, a score 0 (hardly ever use toothpaste) or 1 (usually or always use toothpaste) is given.

CONTACTS AND LOCATIONS:
Overall Officials: Levine Gavel, Principal Investigator — Postgraduate Orthodontics; Valentina Elena Arevalo Cabrera, Principal Investigator — Master Student Oral Health Sciences; Deseyne Thomas, Principal Investigator — Alumnus Orthodontics; Guy AM De Pauw, Study Chair — Professor dr. in Orthodontics; Noëmi MC De Roo, Study Chair — Doctorate in Orthodontics; Liesbeth Temmerman, Study Chair — dr. in Orthodontics
Locations (1):
- University of Ghent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No